CLINICAL TRIAL: NCT02137759
Title: Quantitative Magnetic Resonance Spectroscopic Imaging (MRSI) to Predict Early Response to Standard Radiation Therapy (RT)/Temozolomide (TMZ) ± Belinostat Therapy in Newly-Diagnosed Glioblastomas (GBM)
Brief Title: MRSI to Predict Response to RT/TMZ ± Belinostat in GBM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Emory University (Other)
Collaborators: Johns Hopkins University (Other); Spectrum Pharmaceuticals, Inc (Industry); National Cancer Institute (NCI) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Hui-Kuo Shu, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00065425; Winship2434-13 (Other: Emory Winship Cancer Institute); U01CA172027 (NIH); F30CA206291 (NIH); R21NS100244 (NIH); P30CA138292 (NIH)
Record Dates: First submitted 2014-05-09; First posted 2014-05-14 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Glioblastoma Multiforme of Brain
Keywords: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; belinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Std RT/TMZ (Cohort 1) (Active Comparator): * Standard radiation therapy
  * Standard temozolomide
  Interventions: Radiation: Standard Radiation Therapy; Drug: Standard Temozolomide
- Std RT/TMZ + belinostat (Cohorts 2a, 2b) (Experimental): * Standard radiation therapy
  * Standard temozolomide
  * Belinostat
  Interventions: Radiation: Standard Radiation Therapy; Drug: Standard Temozolomide; Drug: Belinostat

INTERVENTIONS:
Radiation: Standard Radiation Therapy — Radiation therapy to 60 Gy
Drug: Standard Temozolomide — Temozolomide given orally
  Other Names: Temodar
Drug: Belinostat — Belinostat dose to be determined, given intravenously over 30-45 minutes
  Other Names: Beleodaq; PXD101
  Arms: Std RT/TMZ + belinostat (Cohorts 2a, 2b)

SUMMARY:
In the first phase of this study (Cohort 1), the investigators will determine the feasibility of adding MRSI to the evaluation of newly-diagnosed GBM patients treated with standard RT/TMZ and determine whether magnetic resonance spectroscopic imaging (MRSI) can predict for better outcomes in these patients. In the second phase of this study (Cohorts 2a and 2b), the investigators will find the maximum tolerated dose of belinostat for treating newly-diagnosed GBM patients with standard RT/TMZ and will determine whether MRSI can aid clinicians in the early determination of response to this new therapy.

DETAILED DESCRIPTION:
Patients will be assigned to Cohort 1 (standard RT/TMZ) followed by entry to either Cohort 1 or Cohort 2a (standard RT/TMZ + dose finding for belinostat), followed by assignment to Cohort 2b (standard RT/TMZ + tolerable dose of belinostat).

Patients will undergo MRSI scans before beginning treatment and then at several time points during treatment to look for the early response of their tumor to treatment. Blood and tumor samples will be used to measure the levels of certain markers within the cancer cells. Patients will also be assessed for the side effects they experience. Progression-free and overall survival outcomes will be recorded. Patients will also have assessment of their depressive symptoms, quality-of-life and neurocognitive function at several time points during and after therapy course.

ELIGIBILITY:
Inclusion Criteria:

* Newly-diagnosed glioblastoma or gliosarcoma that has been confirmed pathologically
* ≥ 18 years of age
* Able to have MRI scans
* Measurable contrast-enhancing supratentorial tumor (≥ 0.2 cc (current resolution of MRSI is 0.108cc)) in a region amenable to MRSI
* Have the following lab values ≤ 14 days prior to registration:

  * white blood cell count ≥ 3,000/μL
  * absolute neutrophil count ≥ 1,500/μL
  * platelet count of ≥ 100,000/μL
  * hemoglobin ≥ 10 gm/dL (transfusion is allowed to reach minimum level)
  * serum glutamic-oxaloacetic transaminase (SGOT) ≤ 2.0x upper normal limit (UNL)
  * bilirubin ≤ 2 x UNL
  * creatinine ≤ 1.5 mg/dL
* Life expectancy of ≥ 12 weeks
* Karnofsky Performance Score ≥ 60
* Women of childbearing potential must have a negative beta-human chorionic gonadotropin pregnancy test documented ≤ 7 days prior to registration
* All men and women of childbearing potential must agree to use adequate barrier contraception for the duration of study participation and for 12 weeks after the last dose of study drug (If pregnancy or suspected pregnancy occur while participating in study, treating physician should be informed immediately)
* Understand and provide written informed consent
* Both men and women, and members of all races and ethnic groups are eligible for this trial (Subjects will be approximately representative of the demographics of the referral base for the participating institutions)
* Able to swallow capsules
* Willing to provide mandatory tissue samples (unstained slides) for research purposes
* Willing to forego other cytotoxic and non-cytotoxic therapies against the tumor while being treated on this protocol

Exclusion Criteria:

* Pacemakers, non-titanium aneurysm clips, neurostimulators, cochlear implants, non-titanium metal in ocular structures, history of being a steel worker, or other incompatible implants which makes MRI safety an issue
* Any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy
* History of any other invasive cancer (except non-melanoma skin cancer and excluding carcinoma in-situ), unless in complete remission and off of all therapy for that disease for ≥ 3 years, are ineligible
* Active infection or serious intercurrent medical illness
* Any disease that will obscure toxicity or dangerously alter drug metabolism
* Receiving any other investigational agents
* Received prior cytotoxic, non-cytotoxic or experimental drug therapies for brain tumor
* History of prior cranial radiation
* History of myocardial infarction or unstable angina ≤ 6 months prior to registration or congestive heart failure (CHF) requiring use of ongoing maintenance therapy, or life-threatening ventricular arrhythmias
* Patients with congenital long QT syndrome (for cohorts 2a and 2b [belinostat cohorts] only, ECG not required for cohort 1)
* Has prolonged corrected QT (QTc) interval (> 450 msec) (for cohorts 2a and 2b [belinostat cohorts] only, ECG not required for cohort 1)
* Taking any of the following Category I drugs that are generally accepted to have a risk of causing Torsades de Pointes ≤ 7 days prior to registration (for cohorts 2a and 2b [belinostat cohorts] only)

  * Quinidine, procainamide, disopyramide
  * Amiodarone, sotalol, ibutilide, dofetilide
  * Erythromycin, clarithromycin
  * Chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide
  * Cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine
* Taking valproic acid ≤ 2 weeks prior to initiation of belinostat therapy (for cohorts 2a and 2b [belinostat cohorts] only)
* Residual enhancing tumor that lies completely within 1-2 cm of the inner table of the skull (Please consult study neuroradiologist or study PIs at your site if there is uncertainty regarding this exclusion criteria)
* May not be enrolled on any other therapeutic trial for which they are receiving an anti-tumor therapy. (Note: patients on the standard therapy arm of another GBM trial that otherwise meet eligibility requirements for this trial remain eligible for cohort 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-05-07 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) (Cohort 1) | 9 months
  The investigators will use a support vector machine approach to determine an MRSI 5-metabolite profile at week 3 in Cohort 1 that is predictive of prolonged PFS at 9 months.
Maximum Tolerated Dose of Belinostat (Cohort 2a) | 9 weeks
  The investigators will determine the maximum tolerated dose of belinostat (up to 1000 mg/day x 5 days q3weeks x 3) used with standard RT/temozolomide for newly diagnosed GBM patients.
Progression Free Survival (PFS) (Cohort 2b) | 9 months
  The investigators will determine if MRSI biomarkers at week 3 in GBM patients from Cohort 2b can distinguish belinostat responders from non-responders and predict improved PFS at 9 months.

SECONDARY OUTCOMES:
Overall Survival | 18 months
  The investigators will determine whether changes in MRSI metabolite maps at day 8 (for Cohort 2 only), week 3 (for Cohort 1 and 2) and week 11 (for Cohort 1 and 2) predict for overall survival at 18 months.
Progression Free Survival | 9 months
  The investigators will determine whether changes in MRSI metabolite maps at day 8 (for Cohort 2 only) and week 11 (for Cohort 1 and 2) predict for PFS at 9 months.
IDS-SR score change | 11 weeks
  The investigators will determine whether changes in the MRSI metabolite map at week 11 predict for mood alterations as measure by the Inventory of Depressive Symptomatology-Self Report (IDS-SR), a validated instrument for depression assessment, in Cohorts 1 and 2.

OTHER OUTCOMES:
QOL changes | up to 2 years
  The investigators will determine whether changes in MRSI metabolite maps correlate with changes in subjects' quality-of-life (QOL) as measured by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30/Brain Cancer Module-20 (QLQ-C30/BN20) and the MD Anderson Symptom Inventory-Brain Tumor (MDASI-BT), validated instruments for assessing QOL in brain tumor patients.
Neurocognitive function changes | up to 2 years
  The investigators will determine whether changes in MRSI metabolite maps correlate with changes in subjects' neurocognitive function as measured by the Hopkins Verbal Learning Test-Revised (HVLT-R), the Controlled Oral Word Association (COWA) Test and the Trail Making Test (TMT) Parts A & B, validated instruments for evaluating neurocognitive function in brain tumor patients.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Kuo Shu, MD, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT02137759/ICF_001.pdf